CLINICAL TRIAL: NCT04712513
Title: Multicenter Diagnostic Performance of Dynamic CT Perfusion for Functional Assessment of Coronary Artery Disease
Brief Title: Dynamic CT Perfusion for Functional Assessment of Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Aaron So, Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 12052020
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Computed Tomography; Myocardial Perfusion; Fractional Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with coronary artery disease and hemodynamically stable
  Interventions: Diagnostic Test: Dynamic cardiac CT perfusion imaging

INTERVENTIONS:
Diagnostic Test: Dynamic cardiac CT perfusion imaging — Multiple images of the heart are acquired with a clinical CT scanner after an intravenous bolus injection of contrast solution. The images are then analyzed to provide fractional flow reserve and myocardial perfusion values.

SUMMARY:
The objective of this multicenter study is to evaluate the diagnostic accuracy of dynamic cardiac CT perfusion (CTP) imaging for non-invasive functional assessment of coronary artery disease (CAD). The proposed CTP technique allows concomitant assessment of two imaging-derived cardiac biomarkers including fractional flow reserve (FFR) and myocardial perfusion from a single dynamic imaging sequence, which facilities simultaneous evaluation of the hemodynamics in epicardial coronary arteries and coronary microcirculation in patients with CAD. The CTP results will be compared with invasive coronary angiography / FFR assessment and non-invasive cardiac magnetic resonance imaging (CMR) / radionuclide perfusion assessment.

ELIGIBILITY:
1. Subject Inclusion Criteria

   Patients need to meet all the following inclusion criteria to be enrolled in the study:
   1. Symptomatic and hemodynamically stable
   2. Acute coronary syndrome (ACS) ruled out based on absence of abnormal changes in ECG and cardiac enzymes
   3. Referral for cardiac catheterization based on clinical history and non-invasive imaging test findings. Non-invasive imaging findings include one or more of the following: (i) Evidence of myocardial ischemia from radionuclide myocardial perfusion imaging; (ii) Evidence of myocardial ischemia from CMR myocardial perfusion imaging; (iii) Evidence of ≥ 50% stenosis in the left circumflex artery (LCx), left anterior descending artery (LAD) and/or right coronary artery (RCA) from CCTA.
   4. Ability to undergo stress myocardial perfusion test (absence of contraindications for vasodilator)
   5. Written informed consent
2. Subject Exclusion Criteria

Patients meeting at least one of the following criteria will be excluded from the study:

1. Recent (< 1 month) ACS
2. CCTA reveals ≥ 50% stenosis in the left main artery
3. Severe chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
4. Contraindications to stress perfusion imaging, including: i) severe reactive airway disease; ii) high-grade atrioventricular block; iii) allergy to vasodilators; iv) caffeine within 12 hours; v) theophylline use within 48 hours.
5. History of CABG surgery
6. History of malignancy during the past 3 years prior to screening
7. History of alcohol and/or drug abuse within 3 years prior to screening
8. Sign of pregnancy
9. Pregnant or nursing
10. History of severe allergic or anaphylactic reaction to any allergen including drugs and contrast agents
11. Recent (< 1 month) use of an investigational drug or device
12. Participation in any other investigational drug or device trial during the conduct of this study
13. Lack of ability or willingness to comply with the protocol requirements or deemed by the Site Investigator to be unfit for the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are those who have clinically indicated referral for cardiac catheterization based on clinical history and sign of ischemia or obstructive coronary lesion(s) from non-invasive imaging test (radionuclide myocardial perfusion imaging, CMR myocardial perfusion imaging, or CCTA).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of myocardial perfusion obtained from dynamic cardiac CT perfusion imaging for detecting functionally significant coronary artery stenosis | Within 4 weeks prior to invasive cardiac catheterization
  Comparison with invasive coronary angiography and FFR assessment
Accuracy of FFR obtained from dynamic cardiac CT perfusion imaging for detecting functionally significant coronary artery stenosis | Within 4 weeks prior to invasive cardiac catheterization
  Comparison with invasive coronary angiography and FFR assessment
Accuracy of combined myocardial perfusion and FFR measurement obtained from dynamic cardiac CT perfusion imaging for detecting functionally significant coronary artery stenosis | Within 4 weeks prior to invasive cardiac catheterization
  Comparison with invasive coronary angiography and FFR assessment
Comparison of diagnostic accuracy for functional CAD assessment between dynamic CT perfusion and static CT perfusion | Within 4 weeks prior to invasive cardiac catheterization
  Comparison in patients with multi-vessel CAD where balanced ischemia is expected
Comparison of diagnostic accuracy for functional CAD assessment between dynamic CT perfusion and CT-FFR (based on computational fluid dynamics simulation) | Within 4 weeks prior to invasive cardiac catheterization
  Comparison in patients with dense coronary calcification

SECONDARY OUTCOMES:
Comparison of diagnostic accuracy for functional CAD assessment between dynamic CT perfusion and other non-CT perfusion imaging techniques | Within 4 weeks of the acquisition of non-CT perfusion imaging
  Comparison with CMR / radionuclide perfusion assessment
Comparison of diagnostic accuracy of dynamic CT perfusion for functional CAD assessment between male and female patients | Within 4 weeks prior to invasive cardiac catheterization
  Sex-based analysis

CONTACTS AND LOCATIONS:
Locations (1):
- St Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No